CLINICAL TRIAL: NCT00004048
Title: Phase I/II Radioimmunotherapy With High-Dose 90Y-Labeled Humanized MN-14 Alone or Combined With Doxorubicin and Peripheral Blood Stem Cell Rescue (PBSCR) in Medullary Thyroid Cancer (MTC) Grant Application Title: Radioimmunotherapy of MTC With Y-90 Humanized MN14 Anti-CEA Mab and Doxorubicin
Brief Title: Radioimmunotherapy With or Without Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Thyroid Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Garden State Cancer Center at the Center for Molecular Medicine and Immunology (Other)
Responsible Party: Robert M Sharkey, Garden State Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000067172; CMMI-C-040A-98; CMMI-FDR001555; NCI-V99-1564
Record Dates: First submitted 1999-12-10; First posted 2004-04-15 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Head and Neck Cancer
Keywords: thyroid gland medullary carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Medullary | interventions — Filgrastim; Doxorubicin; Peripheral Blood Stem Cell Transplantation; Indium

INTERVENTIONS:
Biological: filgrastim
Drug: doxorubicin hydrochloride
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: indium In 111 monoclonal antibody MN-14
Radiation: yttrium Y 90 monoclonal antibody MN-14

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate tumor cells and deliver tumor-killing substances to them without harming normal cells. Chemotherapy uses different ways to stop tumor cells from dividing so they stop growing or die. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by radioimmunotherapy or chemotherapy used to kill tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of radioimmunotherapy with or without doxorubicin plus peripheral stem cell transplantation in treating patients who have thyroid cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and dose limiting toxicities of high dose yttrium Y 90 monoclonal antibody MN-14 with or without doxorubicin plus peripheral blood stem cell rescue in patients with medullary thyroid cancer. II. Correlate organ and tumor dosimetry with toxicity and antitumor responses in these patients. III. Assess response and duration of response in these patients after this treatment.

OUTLINE: This is a dose escalation study of yttrrium Y 90 monoclonal antibody MN-14 (90Y-MN-14). Patients are stratified by prior doxorubicin (yes vs no). Patients receive filgrastim (G-CSF) subcutaneously (SQ) on days -11 to -7 and undergo leukapheresis on days -8 to -6. If an adequate number of CD34+ cells are not harvested, bone marrow is also collected. Patients receive pretherapy targeting consisting of indium In 111 monoclonal antibody MN-14 (In111-MN-14) on day 0. At least 1 confirmed tumor site must be targeted. Patients receive 90Y-MN-14 IV over 30-45 minutes on day 7. Some patients also receive doxorubicin IV on day 8. PBSC or bone marrow is reinfused on approximately day 7-14. Patients also receive G-CSF SQ or IV until blood counts recover. Cohorts of 3-6 patients receive escalating radiological doses of 90Y-MN-14 until the maximum tolerated dose (MTD) is determined. The MTD is defined as either the dose at which no more than 1 of 6 patients experiences dose limiting toxicity or the threshold radiation doses to lungs, kidneys, and liver. Patients are followed weekly for the first month, monthly for 3 months, then every 6 months for up to 5 years.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for each stratum of this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven medullary thyroid carcinoma Unresectable local-regional disease OR Distant metastases Autologous peripheral blood stem cells (PBSC) or bone marrow available Diffuse bone/marrow involvement allowed if: Autologous bone marrow or PBSC with no greater than 5% tumor involvement available Radiation dose to marrow no greater than 3000 cGy until 6 patients have been treated safely at that dose level At least 1 site confirmed by CT targeted by pretherapy indium In 111 monoclonal antibody MN-14 imaging

PATIENT CHARACTERISTICS: Age: 16 to 80 Performance status: Karnofsky 60-100% ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: WBC at least 3000/mm3 Granulocyte count at least 1500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 mg/dL Renal: Creatinine less than 1.5 times upper limit of normal Cardiovascular: Ejection fraction at least 50% Other: No severe anorexia, nausea, or vomiting No concurrent significant medical complications that would preclude compliance Not pregnant Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since biologic therapy Chemotherapy: At least 4 weeks since prior chemotherapy and recovered No greater than 240 mg/m2 doxorubicin total for combination therapy with doxorubicin but no greater than 550 mg/m2 doxorubicin if radioimmunotherapy alone No prior failure on doxorubicin therapy for combination therapy but not radioimmunotherapy alone Endocrine therapy: Prior synthroid (T4) allowed Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy to index lesion and recovered No prior radiotherapy to greater than 35% of red marrow Surgery: At least 4 weeks since prior major surgery

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1998-09; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack D. Burton, MD, Study Chair — Garden State Cancer Center at the Center for Molecular Medicine and Immunology
Locations (2):
- United States (2):
  - Garden State Cancer Center, Belleville, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey